CLINICAL TRIAL: NCT04707560
Title: Comparison of Heparin-based Wet Suction Method With Dry Suction Method in EUS Fine Needle Biopsy of Solid Pancreatic Mass
Brief Title: Heparin-based Wet Suction Method in EUS Fine Needle Biopsy of Solid Pancreatic Mass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NationalCheng-KungU
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-12

CONDITIONS: Endoscopic Ultrasonography; EUS-FNA; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin Wet first group (Experimental): Heparin based wet suction method of EUS FNB will go first for 2 passes and then shift to dry suction method for another 2 passes.
  Interventions: Procedure: EUS fine needle biopsy with heparin wet suction
- Dry suction first group (Experimental): Dry suction method of EUS FNB will go first for 2 passes and then shift to heparin base wet suction method for another 2 passes.
  Interventions: Procedure: EUS fine needle biopsy with heparin wet suction

INTERVENTIONS:
Procedure: EUS fine needle biopsy with heparin wet suction — EUS FNB with Heparin wet suction:
  Investigator will remove stylet from the FNB device and then infuse Heparin 1ml (5000IU) into device before procedure. The syringe will pre-loaded with 10 ml negative pressure and attach to device upon needle tip insertion into mass lesion.
  EUS FNB with Dry suction:
  Investigator will remove stylet from the FNB device. Syringe will be pre-loaded with 10 ml negative pressure in syringe and attach to needle tail upon needle tip inserted into target lesion.
  Other Names: EUS fine needle biopsy with dry suction

SUMMARY:
The objective of this randomized cross-over trial is to evaluate whether Heparin based wet suction technique, compared with dry suction technique, shall present a higher quality tissue core by using quantitative macroscopic and microscopic scale.

DETAILED DESCRIPTION:
Background & aim Endoscopic ultrasound guided fine needle biopsy (EUS-FNB) is the main tool for tissue acquisition and pathological diagnosis of pancreatic solid mass because of its superior accuracy and lower complication rate compared to CT-guided biopsy. However, the tissue adequacy and diagnostic yield remained unsatisfactory for 2 reasons. First, the conventional dry suction technique (DST) often get small tissue and 3 or more needle passes (i.e. biopsies) are required to obtain enough specimen. Second, blood contamination of the acquired tissue interfered with microscopic examination. Investigator aim to develop a novel technique to improve tissue acquisition within a fewer needle passes and avoid blood contamination by using heparin-based modified wet suction (H-MWST).

Methods This study will be a randomized crossover clinical trial. Patients with pancreatic solid mass indicated for EUS FNB will be enrolled. EUS FNB will be done by one experienced endoscopists in National Cheng Kung University Hospital. Patients will be randomized in a 1:1 ratio to receive EUS FNB with either dry suction technique (DST) or H-MWST first for the initial 2 needle passes, and then crossover to another suction technique for a total of 4 needle passes. The obtained tissue of each needle pass will be sent separately and examined by a pathologist who is unaware of the procedure order. Procedure related complications will be recorded. The primary outcome will be the acquired tissue quality quantified comparison. The secondary outcome will be the overall diagnostic yield, the specimen adequacy, and complication rate by each suction technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients had pancreatic solid mass on CT scan or abdominal echo image

Exclusion Criteria:

* Anti-platelet and anticoagulant user who cannot stop the medication
* Recent acute pancreatitis episode (within 2 weeks)
* Patient with severe cardio-pulmonary dysfunction
* Pregnant women and adolescent < 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of tissue quality | 48 weeks
  White tissue core length will be assessed immediately after procedure. The acquired tumor tissue area and contaminant blood clot percentage will be assessed after total recruitment by single pathologist

SECONDARY OUTCOMES:
Needle pass number needed to establish diagnosis | 48 weeks
  After 5 working days of histology slide preparation and pathologist interpretation. Investigator can get the result
Diagnostic performance between different suction method | 48 weeks
  After 5 working days of histology slide preparation and pathologist interpretation. Investigator can get the result

OTHER OUTCOMES:
Complication | 54 weeks
  Investigator will keep follow up patient during admission course and 3 months after procedure to determine if presented with complications

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Shyang Sheu, Professor, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mok SRS, Diehl DL, Johal AS, Khara HS, Confer BD, Mudireddy PR, Kirchner HL, Chen ZE. A prospective pilot comparison of wet and dry heparinized suction for EUS-guided liver biopsy (with videos). Gastrointest Endosc. 2018 Dec;88(6):919-925. doi: 10.1016/j.gie.2018.07.036. Epub 2018 Aug 16. PMID 30120956
- [Background] Diehl DL, Mok SRS, Khara HS, Johal AS, Kirchner HL, Lin F. Heparin priming of EUS-FNA needles does not adversely affect tissue cytology or immunohistochemical staining. Endosc Int Open. 2018 Mar;6(3):E356-E362. doi: 10.1055/s-0043-121880. Epub 2018 Mar 7. PMID 29527558
- [Background] Kasugai H, Yamamoto R, Tatsuta M, Okano Y, Okuda S, Kishigami Y, Kitamura T, Wada A, Tamura H. Value of heparinized fine-needle aspiration biopsy in liver malignancy. AJR Am J Roentgenol. 1985 Feb;144(2):243-4. doi: 10.2214/ajr.144.2.243. PMID 2981458
- [Background] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Derived] Lin MY, Wu CL, Su YY, Huang CJ, Chang WL, Sheu BS. Tissue Quality Comparison Between Heparinized Wet Suction and Dry Suction in Endoscopic Ultrasound-Fine Needle Biopsy of Solid Pancreatic Masses: A Randomized Crossover Study. Gut Liver. 2023 Mar 15;17(2):318-327. doi: 10.5009/gnl220030. Epub 2022 Sep 2. PMID 36052613